CLINICAL TRIAL: NCT03439553
Title: Estimating the Short-term Effectiveness of Online Advertisements for Improving Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Microsoft Research (Industry)
Collaborators: Schneider Children's Medical Center, Israel (Other); Interdisciplinary Center Herzliya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 177
Record Dates: First submitted 2018-01-31; First posted 2018-02-20 (Actual); Last update posted 2018-02-20 (Actual); Status verified 2018-02

CONDITIONS: Anorexia; Obesity; Smoking Cessation
MeSH Terms: conditions — Anorexia; Obesity; Smoking Cessation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention (Experimental): People shown ads with referral to target websites.
  Interventions: Behavioral: Ads display with target websites
- Intervention with control websites (Active Comparator): People shown ads with referral to control websites.
  Interventions: Behavioral: Ads display with control websites
- Control (No Intervention): People who make target queries, but are not shown the ads.

INTERVENTIONS:
Behavioral: Ads display with target websites — Ads are shown, but users are referred to control websites.
  Arms: Intervention
Behavioral: Ads display with control websites — Ads are shown, but users are referred to control websites.
  Arms: Intervention with control websites

SUMMARY:
Bing ads designed to encourage people to adopt healthier practices (e.g., stop smoking, become physically active, stop consuming harmful content) are shown using the advertising system, to test which ads are more effective as apparent in the subsequent queries to Bing submitted by users who saw the ads.

ELIGIBILITY:
Inclusion Criteria:

* Use of the Bing ad system with target phrases.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2000000 (Actual)
Dates: Start 2015-04-16 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
The number of people who increase and the number of people who decrease searches for positive target behaviors post intervention, compared to prior to the intervention, or a similar decrease in negative behaviors | Up to 1 month after the intervention
  Increase or decrease in searches for positive target behaviors post intervention, compared to prior to the intervention, or a similar decrease in negative behaviors. This measure of outcome was previously used in E. Yom-Tov, Muennig & El-Sayed (2016).

SECONDARY OUTCOMES:
Clickthrough rates | During the intervention itself and up to 1 minute after the intervention (advertisement display).
  Clickthrough rates on each ad

CONTACTS AND LOCATIONS:
Locations (1):
- Microsoft Research Israel, Herzliya, Israel

IPD SHARING:
Plan to Share IPD: No
No IPDs are to be shared with other researchers.

REFERENCES:
- [Derived] Yom-Tov E, Brunstein-Klomek A, Mandel O, Hadas A, Fennig S. Inducing Behavioral Change in Seekers of Pro-Anorexia Content Using Internet Advertisements: Randomized Controlled Trial. JMIR Ment Health. 2018 Feb 22;5(1):e6. doi: 10.2196/mental.8212. PMID 29472176